CLINICAL TRIAL: NCT05788705
Title: Evaluation of the Efficacy of Natural JAK_ STAT Pathways Inhibitors in Treatment of Patients With Rheumatoid Arthritis as a Complementary Medicine
Brief Title: Efficacy of JAK STAT Pathways Inhibitors in Treatment of Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adel A.Gomaa (Other)
Responsible Party: Sponsor-Investigator, Adel A.Gomaa, PROF OF CLINICAL PHARMACOLOGY, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Natural JAK STAT Inhibitors
Record Dates: First submitted 2023-02-27; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Apigenin; Glycyrrhizic Acid; boswellic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "apigenin" and "glycyrrhizin" (Active Comparator): Patients will receive one capsule contains 10 mg of apigenin (Matricaria chamomilla L extract) and one capsule contains glycyrrhizin 50(licorice extract) twice daily for 6 months
  Interventions: Dietary Supplement: "apigenin" and "glycyrrhizin"
- "boswellic acid" and "glycyrrhizin" (Active Comparator): Patients will receive one capsule contains 200 mg boswellic acid (Boswellia serrata extract) and one capsule contains glycyrrhizin 50(licorice extract) twice daily for 6 months
  Interventions: Dietary Supplement: "glycyrrhizin" and "boswellic acid"
- "placebo" (Placebo Comparator): Patients will receive daily two capsules contain placebo for 6 months
  Interventions: Dietary Supplement: "placebo"

INTERVENTIONS:
Dietary Supplement: "apigenin" and "glycyrrhizin" — "apigenin" will be administered as capsule (10mg,eq 200mg Matricaria chamomilla L extract) two times daily. Also, "glycyrrhizin " will be administered as capsule(50 mg eq 250 mg licorice extract) two times daily. The two types of capsules administration will be continue for 6 months
  Arms: "apigenin" and "glycyrrhizin"
Dietary Supplement: "glycyrrhizin" and "boswellic acid" — "boswellic acid" will be administered as capsule (200mg,eq 250mg Boswellia serrata extract) two times daily. Also, "glycyrrhizin " will be administered as capsule(50 mg eq 250 mg licorice extract) two times daily. The two types of capsules administration will be continue for 6 months
  Arms: "boswellic acid" and "glycyrrhizin"
Dietary Supplement: "placebo" — "Placebo "capsule will be administered two times daily for 6 months
  Arms: "placebo"

SUMMARY:
There is no treatment that could utterly cure Rheumatoid arthritis (RA), but the disease is mainly improved by conventional disease-modifying anti rheumatic drugs. Methotrexate and biological DMARDs as JAK-STAT inhibitors may be used to control and delay the progression of the disease and improve the quality of lives of patients. However, DMARDs have deleterious effects on human health. Several natural components have JAK-STAT inhibitory effect such as Boswellic acid (Boswellia serrata extract), Glycyrrhizin (Glycyrrhiza glabra extr.) and Apigenin (Chamomile extr)

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic chronic, progressive, autoimmune disease characterized by inflammatory cell infiltration and synovial proliferation, accompanied by injury to articular cartilage and subchondral bone The prevalence of RA in women is 3.6% and 1.7% for men . There is no treatment that could utterly cure RA, but the disease is mainly improved by conventional disease-modifying antirheumatic drugs. Methotrexate and biological DMARDs as JAK-STAT inhibitors may be used to control and delay the progression of the disease and improve the quality of lives of patients. However, DMARDs have deleterious effects on human health. Chronic use of these agents by pregnant patients may induce teratogenic effects . Many studies showed that some natural plant extracts or mixed herbal compounds effectively regulate the immune system and possess in vitro and/or in vivo inhibitory effects against STAT to alleviate RA by inhibiting pro-inflammatory cytokines. Several natural components have JAK-STAT inhibitory effect such as Boswellic acid (Boswellia serrata extract), Glycyrrhizin (Glycyrrhiza glabra extr.) and Apigenin (Chamomile extr.). Boswellic acid and its derivative acetyl-11- keto boswellic acid, are reported to be the most potent inhibitors in the synthesis of 5-LOX. Since 5-LOX is an important enzyme involved in the biosynthesis of leukotrienes and is significantly expressed in RA. B. serrata extract, when administered orally, inhibits IL-6, IL-1 , IFN- TNF- and PGE2 in complete Freund's adjuvant-induced arthritis in rats. Glycyrrhizin reduced the activity of JAK/STAT signaling pathway, which is the upstream regulator of HMGB1. These natural products have inhibitory effect for the STAT3 signaling pathway that have anti-inflammatory and anti-rheumatoid as well as anticancer effects. These inhibitors have been found to inhibit the STAT3 signaling pathway by reducing IL-6 production . Apigenin is a plant-derived flavonoid that is abundant in celery, Chamomile, plantain seed, and is effective in the prevention and treatment of inflammatory diseases, prostate cancer, and in inhibiting tumorigenesis and angiogenesis in melanoma, breast, skin, and colon cancers. Apigenin reduced p-JAK1/2 and p-STAT3 in breast cancer (BT-474) cells, and demonstrated antirheumatic and anticancer activity by inhibiting JAK-STAT . our aim To assess the efficacy of some natural JAK-STAT inhibitors as complementary medicine in the treatment of rheumatoid arthritis and attenuation of the side effects of regular methotrexate our Research outcome measures:

1. Primary (main):

   1. The change in DAS28 based on C-reactive protein (DAS28-CRP) and the Clinical Disease Activity Index (CDAI)
   2. Rate of achieving 20%, 50% and 70% improvement in the American College Rheumatology criteria (ACR20, ACR50, ACR70).
2. Secondary (subsidiary):

   1. Change in visual analogue scale (VAS).
   2. Determination of effusion synovitis volume on musculoskeletal ultrasound(MSUS)
   3. Determination of Inflammatory cytokines levels: (Tumour necrosis factor α and Interleukin 6).
   4. Safety and Tolerability Measures: adverse events including nausea, vomiting, dizziness and abdominal pain, CBC and urine analysis as well as kidney and liver function tests will be performed before enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,ages18-60.
* Patients who met criteria for the diagnosis of RA
* Patients who were signed the informed consent form.

Exclusion Criteria:

* Patients with Malignant tumours,
* Patients with Infectious diseases,
* Patients with Hematologic diseases.
* Patients with other rheumatic diseases.
* Women who are pregnant or breastfeeding.

  * Hypersensitivity to dietary supplement used in this study.
  * Hypertensive patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The change in DAS28 based on C-reactive protein (DAS28-CRP) | Before the intervention, 3 months after the intervention, and 6 months after the intervention
  DAS-28 score: a DAS-28 score > 5.1 indicating high disease activity; 3.2< DAS-28 score≤5.1 indicates moderate disease activity; 2.6< DAS-28 score≤3.2 indicates low disease activity; DAS-28 score≤2.6 indicates basic disease remission

SECONDARY OUTCOMES:
Change in visual analogue scale (VAS | Before the intervention, 3 months after the intervention, and 6 months after the intervention
  each patient will be asked to indicate his or her current level of pain on 100mm scale.0scale indicate no pain and 100mm indicate worst pain imaginable
Determination of effusion synovitis volume on musculoskeletal ultrasound(MSUS) | Before the intervention, 3 months after the intervention, and 6 months after the intervention
  Determination of effusion synovitis volume on musculoskeletal ultrasound
Determination of Inflammatory cytokines levels: (Tumour necrosis factor α and Interleukin 6). | Before the intervention, 3 months after the intervention, and 6 months after the intervention
  laboratory test

IPD SHARING:
Plan to Share IPD: Yes
Data will become available to interested investigators upon submitting a reasonable research request by email to A. Gomaa
  (a.gomma@aun.edu.eg).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July, 2025
Access Criteria: Data will become available to interested investigators upon submitting a reasonable research request by email to A. Gomaa
  (a.gomma@aun.edu.eg).

REFERENCES:
- [Background] Smolen JS, Aletaha D, McInnes IB. Rheumatoid arthritis. Lancet. 2016 Oct 22;388(10055):2023-2038. doi: 10.1016/S0140-6736(16)30173-8. Epub 2016 May 3. PMID 27156434
- [Background] Guo Q, Wang Y, Xu D, Nossent J, Pavlos NJ, Xu J. Rheumatoid arthritis: pathological mechanisms and modern pharmacologic therapies. Bone Res. 2018 Apr 27;6:15. doi: 10.1038/s41413-018-0016-9. eCollection 2018. PMID 29736302
- [Background] Oton T, Carmona L. The epidemiology of established rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2019 Oct;33(5):101477. doi: 10.1016/j.berh.2019.101477. Epub 2020 Jan 25. PMID 31987685
- [Background] Ytterberg SR, Bhatt DL, Mikuls TR, Koch GG, Fleischmann R, Rivas JL, Germino R, Menon S, Sun Y, Wang C, Shapiro AB, Kanik KS, Connell CA; ORAL Surveillance Investigators. Cardiovascular and Cancer Risk with Tofacitinib in Rheumatoid Arthritis. N Engl J Med. 2022 Jan 27;386(4):316-326. doi: 10.1056/NEJMoa2109927. PMID 35081280
- [Background] Hoisnard L, Pina Vegas L, Dray-Spira R, Weill A, Zureik M, Sbidian E. Risk of major adverse cardiovascular and venous thromboembolism events in patients with rheumatoid arthritis exposed to JAK inhibitors versus adalimumab: a nationwide cohort study. Ann Rheum Dis. 2023 Feb;82(2):182-188. doi: 10.1136/ard-2022-222824. Epub 2022 Oct 5. PMID 36198438
- [Background] Yang J, Wang L, Guan X, Qin JJ. Inhibiting STAT3 signaling pathway by natural products for cancer prevention and therapy: In vitro and in vivo activity and mechanisms of action. Pharmacol Res. 2022 Aug;182:106357. doi: 10.1016/j.phrs.2022.106357. Epub 2022 Jul 19. PMID 35868477
- [Background] Dudics S, Langan D, Meka RR, Venkatesha SH, Berman BM, Che CT, Moudgil KD. Natural Products for the Treatment of Autoimmune Arthritis: Their Mechanisms of Action, Targeted Delivery, and Interplay with the Host Microbiome. Int J Mol Sci. 2018 Aug 24;19(9):2508. doi: 10.3390/ijms19092508. PMID 30149545
- [Background] Kumar R, Singh S, Saksena AK, Pal R, Jaiswal R, Kumar R. Effect of Boswellia Serrata Extract on Acute Inflammatory Parameters and Tumor Necrosis Factor-alpha in Complete Freund's Adjuvant-Induced Animal Model of Rheumatoid Arthritis. Int J Appl Basic Med Res. 2019 Apr-Jun;9(2):100-106. doi: 10.4103/ijabmr.IJABMR_248_18. PMID 31041173
- [Background] Wu X, Wang W, Chen Y, Liu X, Wang J, Qin X, Yuan D, Yu T, Chen G, Mi Y, Mou J, Cui J, Hu A, E Y, Pei D. Glycyrrhizin Suppresses the Growth of Human NSCLC Cell Line HCC827 by Downregulating HMGB1 Level. Biomed Res Int. 2018 Jan 15;2018:6916797. doi: 10.1155/2018/6916797. eCollection 2018. PMID 29568761
- [Background] Wu Y, Wang Z, Du Q, Zhu Z, Chen T, Xue Y, Wang Y, Zeng Q, Shen C, Jiang C, Liu L, Zhu H, Liu Q. Pharmacological Effects and Underlying Mechanisms of Licorice-Derived Flavonoids. Evid Based Complement Alternat Med. 2022 Jan 17;2022:9523071. doi: 10.1155/2022/9523071. eCollection 2022. PMID 35082907
- [Background] Abid R, Ghazanfar S, Farid A, Sulaman SM, Idrees M, Amen RA, Muzammal M, Shahzad MK, Mohamed MO, Khaled AA, Safir W, Ghori I, Elasbali AM, Alharbi B. Pharmacological Properties of 4', 5, 7-Trihydroxyflavone (Apigenin) and Its Impact on Cell Signaling Pathways. Molecules. 2022 Jul 4;27(13):4304. doi: 10.3390/molecules27134304. PMID 35807549